CLINICAL TRIAL: NCT04079049
Title: Breast Cancer Liver Metastases-2 - A Multicentre Randomized Clinical Trial Investigating Local Treatment for Breast Cancer Liver Metastases
Brief Title: BreCLIM-2 - A RCT Investigating Local Treatment for Breast Cancer Liver Metastases
Acronym: BreCLIM-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Uppsala University (Other); Karolinska Institutet (Other); Linkoeping University (Other Government); Lund University (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BreCLIM-2018-116-31M
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Liver Metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical intervention (Experimental): Surgical and oncological treatment
  Interventions: Procedure: Surgical intervention
- Control (Active Comparator): Oncological treatment
  Interventions: Drug: Control

INTERVENTIONS:
Procedure: Surgical intervention — Surgical intervention by liver resection, ablation or stereotactic body radiotherapy as complement to oncological treatment
  Arms: Surgical intervention
Drug: Control — Oncological treatment in control group
  Arms: Control

SUMMARY:
Breast cancer is the second most common cancer in Sweden with an incidence of 8000 per year. The role of surgery for distant breast cancer metastasis beyond local lymph nodes remains controversial even though some reports suggest there might be a survival benefit from resection of oligometastases in the liver.

The purpose of this multicentre randomized clinical trial is to evaluate local treatment for breast cancer liver metastases, compared to systemic oncological treatment only. The primary endpoint is time to death from any cause, which will be compared using cox proportional hazard regression. The secondary endpoints are three years survival, progression-free survival, median overall survival and quality of life. The aim is also to evaluate overall safety and predictive factors for survival during oncological and surgical treatment. The overall purpose is to ameliorate treatment for advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* >18 years old
* ECOG 0-1
* Breast cancer history
* Breast cancer liver metastasis verified by biopsy
* Patient amendable for liver surgery and pre- and postoperative oncological treatment
* 1-4 liver metastasis amendable to surgery with functional liver remnant volume >30%
* Liver metastasis (and skeletal metastasis) stable or responding to preoperative oncological treatment

Exclusion Criteria:

* Non-skeletal extrahepatic disease
* Non-resected primary tumour
* Pregnancy
* Progression of disease upon oncological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Three years after randomization
  Time to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Hemmingsson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden